CLINICAL TRIAL: NCT00401479
Title: An Exploratory Phase I Study in Healthy Volunteers of GI Transit Following Administration of the ß3-Adrenergic Receptor Agonist, Solabegron (Study B3I106248)
Brief Title: A Study To Investigate The Effect Of Solabegron (GW427353) On Gastrointestinal Transit In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: B3I106248
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: GW427353; b3-Adrenergic Receptor Agonist; Irritable Bowel Syndrome (IBS); pharmacokinetics; tolerability; gastrointestinal transit
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — solabegron

INTERVENTIONS:
Drug: Placebo
Drug: Solabegron (GW427353)
  Other Names: Placebo

SUMMARY:
This study will test the hypothesis that GW427353, a beta-3 adrenergic agonist, retards the emptying of the colon and increases total colonic transit time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no evidence of current or past history suggestive of gastrointestinal disease or disorder or medical illness that could compromise interpretation of the study.
* no clinically significant laboratory results collected at the screening visit
* men: body weight greater than or equal to 50kg (110 lbs)
* women: body weight greater than or equal to 45kg (100 lbs)
* BMI between 18.5 - 35 kg/m2

Exclusion Criteria:

* Females who are nursing or pregnant.
* history of inflammatory bowel disease
* history of gastric ulcers within 12 months of signing the informed consent form
* tobacco users

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10

PRIMARY OUTCOMES:
colonic emptying rate by radiolabeled scintigraphy | throughout the study

SECONDARY OUTCOMES:
Safety and tolerability: ECG, vital signs, adverse events, clinical lab tests. Diary card collection of stool frequency Stool consistency and ease of passage Blood levels of GW427353 | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Rochester, Minnesota, United States